CLINICAL TRIAL: NCT01973114
Title: A Randomized, Double Blind, Placebo-controlled, Parallel Group Study to Determine the Efficacy, the Duration of Action, and Safety of Latanoprost in Patients With Menière's Disease
Brief Title: Latanoprost for the Treatment of Menière's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Synphora AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M 05 - 2013
Record Dates: First submitted 2013-10-17; First posted 2013-10-31 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Menière's Disease
Keywords: Menière's disease; Vertigo; Hearing loss; Tinnitus
MeSH Terms: conditions — Vertigo; Hearing Loss; Tinnitus | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Group 1 (Experimental): One intratympanic injection of latanoprost (Day1)
  Interventions: Drug: Latanoprost
- Group 2 (Placebo Comparator): One intratympanic injection of placebo
  Interventions: Other: Placebo
- Group 3 (Experimental): Three intratympanic injections of latanoprost (Day 1, 2 and 3)
  Interventions: Drug: Latanoprost
- Group 4 (Placebo Comparator): Three intratympanic injections of placebo (Day 1, 2 and 3)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Latanoprost
  Arms: Group 1; Group 3
Other: Placebo
  Arms: Group 2; Group 4

SUMMARY:
The purpose of the study is to evaluate the dose regimen, efficacy and safety of latanoprost for the treatment of Menière's disease.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Definitive unilateral Menière's disease (AAO-HNS 1995)
* Disease stage II - III: PTA4 (Pure Tone Average) (0.5, 1.0, 2.0 and 3.0kHz) between 25dB and 70dB
* Speech discrimination score in silence: No better than 85%
* At least three vertigo attacks (lasting ≥ 20 minutes) during the last three months prior to inclusion
* Tinnitus during the last three months prior to inclusion
* Signed written informed consent

Exclusion Criteria:

* Medical or psychiatric conditions which could jeopardize or would compromise the subject's ability to participate in the trial or decrease the likelihood of obtaining satisfactory data to achieve the objective of the trial, dementia, alcohol or substance abuse.
* Bilateral Menière's disease
* Chronic otitis media on the ear affected by Menière's disease
* Subjects not fluent in Swedish language
* Bronchial asthma
* Previous intratympanic injection of gentamicin or surgical therapy
* Previous intratympanic steroid therapy less than six months prior to inclusion
* Known hypersensitivity to local anesthetics
* Pregnant women
* Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change in speech discrimination score in noise from Baseline | 2 weeks

SECONDARY OUTCOMES:
Change in speech discrimination score in noise from Baseline | 3 months
Change in pure tone audiometry from Baseline | 3 months
Change in THI-25 (Tinnitus Handicap Inventory) score from Baseline | 3 months
Change in hearing (Likert scale), tinnitus (Likert scale) and vertigo (Likert scale) from run-in period | 3 months
Change in proportion of days with vertigo attacks from run-in period | 3 months
Comparison of number of drop attacks in each treatment arm | 3 months
Evaluation of adverse events and vital signs as measure of safety and tolerability | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Karlberg, MD, PhD, Principal Investigator — Lund University Hospital
Locations (12):
- Sweden (12):
  - Falu Lasarett, Falun
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Blekinge Hospital, Karlskrona
  - Centralsjukhuset i Karlstad, Karlstad
  - Centralsjukhuset i Kristianstad, Kristianstad
  - Linköping University Hospital, Linköping
  - Sunderby Sjukhus, Luleå
  - Lund University Hospital, Lund
  - University Hospital Örebro, Örebro
  - Karolinska Universitetssjukhuset, Stockholm
  - Uppsala University Hospital, Uppsala
  - Västmanlands Sjukhus i Västerås, Västerås